CLINICAL TRIAL: NCT05684796
Title: STORM-PE: A Prospective, Multicenter, Randomized Controlled Trial Evaluating Anticoagulation Alone vs Anticoagulation Plus Mechanical Aspiration With the Indigo® Aspiration System for the Treatment of Intermediate High Risk Acute Pulmonary Embolism
Brief Title: Comparison of Two Pulmonary Embolism Treatments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penumbra Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18190
Record Dates: First submitted 2022-12-16; First posted 2023-01-13 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Pulmonary Embolism Acute
Keywords: intermediate-high risk; acute; PE; clot

STUDY DESIGN:
Intervention Model Description: Randomization will be 1:1 to either anticoagulation alone (AC Group) or anticoagulation plus mechanical aspiration thrombectomy with the Indigo Aspiration System (Indigo Group).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Anticoagulation (AC) (Active Comparator): Subjects will have their pulmonary embolism treated with anticoagulants alone. There will be no procedure for this group.
  Interventions: Drug: Anticoagulation
- Indigo (Active Comparator): Subjects will have their pulmonary embolism treated with anticoagulants and mechanical aspiration thrombectomy with the Indigo® Aspiration System.
  Interventions: Device: mechanical aspiration thrombectomy

INTERVENTIONS:
Drug: Anticoagulation — Anticoagulation with unfractionated heparin (UFH) or low molecular weight heparin (LMWH)
  Arms: Anticoagulation (AC)
Device: mechanical aspiration thrombectomy — Mechanical aspiration thrombectomy with the Indigo Aspiration System.
  Other Names: Indigo Aspiration System
  Arms: Indigo

SUMMARY:
The primary objective of this trial is to evaluate the safety and efficacy of treatment with anticoagulation alone versus anticoagulation and mechanical aspiration thrombectomy with the Indigo Aspiration System for the treatment of intermediate-high risk acute pulmonary embolism (PE).

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years old
2. Clinical signs and symptoms consistent with acute PE with duration of 14 days or less
3. Objectively confirmed acute PE, based on computed tomographic pulmonary angiography (CTPA) imaging showing a filling defect in at least one main or proximal lobar pulmonary artery
4. Classification of intermediate high-risk PE as demonstrated by right ventricular dysfunction with RV/LV ratio ≥1.0 on CTPA and elevated cardiac biomarkers, including cardiac troponin, BNP, and/or NT-pro BNP above the upper limit of normal
5. Jugular or femoral access deemed suitable to accommodate pulmonary artery intervention with the Indigo Aspiration System
6. Informed consent is obtained from either the patient or legally authorized representative (LAR)

Exclusion Criteria:

1. Administration of thrombolytic agents or glycoprotein IIb/IIIa receptor antagonist within 30 days prior to baseline imaging
2. Hemodynamic instability with any of the following present:

   1. Cardiac arrest
   2. Obstructive shock or persistent hypotension defined as systolic blood pressure (BP) <90 mmHg or an acute drop in systolic BP ≥40 mmHg for >15 min, or requiring vasopressor or inotropic support to achieve a systolic BP ≥90 mmHg
3. Patients on ECMO
4. National Early Warning Score (NEWS) 2 ≥9
5. History, imaging or hemodynamic findings consistent with chronic thromboembolic pulmonary hypertension (CTEPH) or chronic thromboembolic disease (CTED) diagnosis
6. Imaging evidence or other evidence that suggests, in the opinion of the Investigator, that catheter-based intervention is not appropriate for the patient
7. Allergy, hypersensitivity, or heparin induced thrombocytopenia (HIT)
8. Contraindication or sensitivity to iodinated intravascular contrast that cannot be adequately premedicated
9. <45 mL/min creatinine clearance
10. Severe active infection (e.g. sepsis) requiring treatment at time of enrollment
11. Active bleeding or disorders contraindicating anticoagulant therapy
12. Hemoglobin <10 g/dL
13. Platelets <100,000/μL
14. INR >3
15. Cardiovascular or pulmonary surgery within last 7 days
16. Primary brain or metastatic brain cancer
17. Life expectancy <90 days
18. Pregnancy
19. Intracardiac thrombus (right atrium, right ventricle clot in transit) or thrombus in the inferior vena cava identified on baseline imaging
20. Current participation in another investigational drug or device trial that may confound the results of this trial. Studies requiring extended follow-up for products that were investigational but have since become commercially available are not considered investigational studies.
21. Other medical, social, or psychological conditions that, in the opinion of the Investigator, precludes the patient from appropriate consent, could limit the patient's ability to participate in the trial, including compliance with follow-up requirements, or that could impact the scientific integrity of the trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-11-27 (Actual); Primary Completion 2025-06-12 (Actual); Study Completion 2025-09-09 (Actual)

PRIMARY OUTCOMES:
Change in RV/LV ratio | 48 hours post-randomization
  Change in RV/LV ratio at 48 hours on original therapy as assessed by computerized tomography pulmonary angiogram (CTPA)

SECONDARY OUTCOMES:
Major Adverse Events | within 7 days post-randomization
  Major adverse events (MAEs) within 7 days: a composite of clinical deterioration requiring escalation of care, PE-related mortality, symptomatic recurrent PE, or major bleeding
Functional Outcome Assessment with the 6-minute walk test | within 90 days post-randomization
  Functional outcome as assessed by the 6-minute walk test (6MWT) through 90 days. The 6-minute walk test measures distance walked in meters, with longer distances being better.
Functional Outcome Assessment with the New York Heart Association Classification | within 90 days post-randomization
  Functional outcome as assessed by the New York Heart Association classification (NYHA) through 90 days. The New York Heart Association classification ranges from Class I-IV, with higher classifications being worse.
Functional Outcome Assessment with the Post Venous Thromboembolism Functional Status scale | within 90 days post-randomization
  Functional outcome as assessed by the Post Venous Thromboembolism Functional Status (PVFS) scale through 90 days. The Post Venous Thromboembolism Functional Status scale ranges from 0-5, with higher scores being worse.
Functional Outcome Assessment with the modified Medical Research Council Dyspnea Scale | within 90 days post-randomization
  Functional outcome as assessed by the modified Medical Research Council Dyspnea Scale (mMRC) through 90 days. The modified Medical Research Council Dyspnea Scale ranges from 0-4, with higher scores being worse.
Functional Outcome Assessment with the Borg Scale | within 90 days post-randomization
  Functional outcome as assessed by the Borg Scale through 90 days. The Borg Scale ranges from 0-10, with higher scores being worse.
Quality of Life Assessment with the Pulmonary Embolism Quality of Life Questionnaire | within 90 days post-randomization
  Quality of Life (QoL), as assessed by the Pulmonary Embolism Quality of Life Questionnaire (PEmb-QoL) through 90 days. The Pulmonary Embolism Quality of Life Questionnaire measures 6 dimensions, with higher scores being worse.
Quality of Life Assessment with the EQ-5D-5L Questionnaire | within 90 days post-randomization
  Quality of Life (QoL), as assessed by the EQ-5D-5L Questionnaire through 90 days. The EQ-5D-5L Questionnaire measures 5 dimensions, with higher scores being worse.
  The Visual Analogue Scale (VAS) scale is part of the questionnaire and ranges from 0-100, with higher scores being better.
All-cause Mortality | within 90 days post-randomization
  All-cause mortality within 90 days
PE-related Mortality | within 90 days post-randomization
  PE-related mortality within 90 days
Symptomatic PE Recurrence | within 90 days post-randomization
  Symptomatic PE recurrence within 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Rosovsky, MD, Principal Investigator — Massachusetts General Hospital; Robert Lookstein, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (22):
- United States (19):
  - The University of Arizona - Banner, Tucson, Arizona
  - UCLA Medical Center, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Radiology and Imaging Specialists/Lakeland Regional, Lakeland, Florida
  - Joseph Maxwell Cleland Atlanta VA Medical Center, Decatur, Georgia
  - Wellstar Kennestone, Marietta, Georgia
  - Northwestern Memorial, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - St. Elizabeth Edgewood Hospital, Edgewood, Kentucky
  - University of Maryland, Baltimore, Maryland
  - McLaren Bay Heart & Vascular, Bay City, Michigan
  - Corewell Health William Beaumont University Hospital, Royal Oak, Michigan
  - Cooper Health System, Camden, New Jersey
  - Mount Sinai Hospital, New York, New York
  - Ascension Seton Medical Center Austin, Austin, Texas
  - Baylor University Medical Center, Dallas, Texas
  - Kingwood Medical Center, Kingwood, Texas
  - Metropolitan Methodist Hospital, San Antonio, Texas
  - Sentara Norfolk General Hospital, Norfolk, Virginia
- Foothills Medical Centre, Calgary, Alberta, Canada
- Auckland City Hospital, Auckland, New Zealand
- Krakowski Szpital Specjalistyczny św. Jana Pawła II, Krakow, Poland

REFERENCES:
- [Derived] Lookstein RA, Konstantinides SV, Weinberg I, Dohad SY, Rosol Z, Kopec G, Moriarty JM, Parikh SA, Holden A, Channick RN, McDonald B, Nagarsheth KH, Yamada K, Rosovsky RP; STORM-PE Trial Investigators. Randomized Controlled Trial of Mechanical Thrombectomy With Anticoagulation Versus Anticoagulation Alone for Acute Intermediate-High Risk Pulmonary Embolism: Primary Outcomes From the STORM-PE Trial. Circulation. 2026 Jan 6;153(1):21-34. doi: 10.1161/CIRCULATIONAHA.125.077232. Epub 2025 Nov 3. PMID 41183181
- [Derived] Rosovsky RP, Konstantinides SV, Moriarty JM, Dohad SY, Weinberg I, Parikh SA, Channick R, Lookstein RA. A prospective, multicenter, randomized controlled trial evaluating anticoagulation alone vs anticoagulation plus computer assisted vacuum thrombectomy for the treatment of intermediate-high-risk acute pulmonary embolism: Rationale and design of the STORM-PE study. Am Heart J. 2025 Oct;288:1-14. doi: 10.1016/j.ahj.2025.03.018. Epub 2025 Mar 31. PMID 40174693